CLINICAL TRIAL: NCT01764789
Title: A Biobehavioral Intervention for Patients With Gynecologic or Breast Cancer Recurrence
Brief Title: Stress Reduction in Improving Quality of Life in Patients With Recurrent Gynecologic or Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Barbara Andersen, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: OSU-10026; NCI-2012-01177 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); R21CA135005 (NIH)
Record Dates: First submitted 2013-01-08; First posted 2013-01-10 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2015-10

CONDITIONS: Anxiety Disorder; Depression; Fatigue; Leydig Cell Tumor; Ovarian Sarcoma; Ovarian Stromal Cancer; Pain; Peritoneal Carcinomatosis; Pseudomyxoma Peritonei; Recurrent Breast Cancer; Recurrent Cervical Cancer; Recurrent Endometrial Carcinoma; Recurrent Fallopian Tube Cancer; Recurrent Gestational Trophoblastic Tumor; Recurrent Ovarian Epithelial Cancer; Recurrent Ovarian Germ Cell Tumor; Recurrent Primary Peritoneal Cavity Cancer; Recurrent Uterine Sarcoma; Recurrent Vaginal Cancer; Recurrent Vulvar Cancer
Keywords: psychological intervention; breast cancer; gynecologic cancer
MeSH Terms: conditions — Anxiety Disorders; Depression; Fatigue; Leydig Cell Tumor; Pain; Peritoneal Neoplasms; Pseudomyxoma Peritonei; Breast Neoplasms; Uterine Cervical Neoplasms; Endometrial Neoplasms; Fallopian Tube Neoplasms; Gestational Trophoblastic Disease; Carcinoma, Ovarian Epithelial; Vaginal Neoplasms; Vulvar Neoplasms | interventions — Psychiatric Rehabilitation; Behavior Therapy; Early Intervention, Educational; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Supportive care (psychosocial intervention) (Experimental): Patients participate in a multi-component intervention based on cognitive and behavioral principles comprising MBSR, an intervention to promote hopefulness, and a problem solving approach which navigates around obstacles or generates alternatives when goals become blocked. Additional topics may be covered as indicated by clinical need and patients goals. Biobehavioral components include addressing social and disease-specific quality of life, and pain education. Intensive treatment sessions continue weekly for 16 weeks followed by 2 biweekly and 2 monthly maintenance sessions.
  Interventions: Other: questionnaire administration; Procedure: quality-of-life assessment; Procedure: psychosocial assessment and care; Behavioral: behavioral intervention; Other: cognitive intervention; Other: educational intervention

INTERVENTIONS:
Other: questionnaire administration — Ancillary studies
Procedure: quality-of-life assessment — Patients will participate in a quality life assessment.
  Other Names: quality of life assessment; Ancillary studies
Procedure: psychosocial assessment and care — Participate in multi-component biobehavioral intervention
  Other Names: psychosocial assessment; psychosocial assessment/care; psychosocial care; psychosocial care/assessment; psychosocial studies
Behavioral: behavioral intervention — Participate in multi-component biobehavioral intervention
  Other Names: Behavior Conditioning Therapy; Behavior Therapy; Behavioral Modification; Behavioral Therapy; Behavioral Treatment
Other: cognitive intervention — A multi-component intervention based on cognitive and behavioral principles will be used. It combines effective intervention strategies selected for their relevance to patients with recurrent cancer.
Other: educational intervention — Participate in multi-component biobehavioral intervention
  Other Names: intervention, educational

SUMMARY:
This pilot clinical trial studies stress reduction in improving quality of life in patients with recurrent gynecologic or breast cancer. Participating in a stress reduction program may help improve quality of life in patients with gynecologic or breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To refine the intervention. II. Test the acceptability, feasibility, and clinical appropriateness of the intervention.

III. To provide a preliminary test of its efficacy.

OUTLINE:

Patients participate in a multi-component intervention based on cognitive and behavioral principles comprising mindfulness-based stress reduction (MBSR), an intervention to promote hopefulness, and a problem solving approach which navigates around obstacles or generates alternatives when goals become blocked. Additional topics may be covered as indicated by clinical need and patients goals. Biobehavioral components include addressing social and disease-specific quality of life, and pain education. Intensive treatment sessions continue weekly for 16 weeks followed by 2 biweekly and 2 monthly maintenance sessions.

After completion of study treatment, patients are followed up at 28 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of recurrent breast or gynecologic cancer (any site) with any disease-free interval; second primary cancers do not meet this criterion
* English speaking
* Able and willing to give informed consent
* To be considered for the blood and saliva collection, women must fulfill the following secondary criteria:

  * Diagnosis of recurrent breast or ovarian cancer with any disease-free interval

Exclusion Criteria:

* Residence > 70 miles from research site
* Subnormal intellectual potential (diagnosis of mental retardation)
* Progressive neurological or chronic, progressive, debilitating condition (e.g., dementia)
* Non-ambulatory
* Life expectancy less than 160 days, per the treating oncologist
* Current suicide risk sufficient to preclude treatment on an outpatient basis
* Chronic inflammatory or autoimmune disorder (e.g., rheumatoid arthritis, lupus)

Ages: 21 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2010-10; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Quality of life(QoL) | up to 28 weeks
  Quality of life as assessed by Short Form (SF)-36

SECONDARY OUTCOMES:
Mood as assessed by the Profile of Mood States (POMS) | Up to 28 weeks
Depressive symptoms as assessed by the Center for Epidemiological Studies, Depression scale (CES-D) | Up to 28 weeks
Stress as assessed by the Impact of Event Scale (IES) | Up to 28 weeks
Pain as assessed by the Brief Pain Inventory (BPI) | Up to 28 weeks
Fatigue as assessed by the Fatigue Severity Index (FSI) | Up to 28 weeks
Diurnal cortisol slope | Up to 28 weeks
  Study participants will also collect saliva samples at home 4 times a day for 3 days. Saliva samples will be collected at the baseline, mid-treatment, post-treatment and 3-month follow-up assessments. These samples will be used to measure cortisol.
Inflammation | Up to 28 weeks
  Blood samples will be used to measure levels of inflammatory markers. Blood draws will be coordinated with the participants' regularly scheduled blood draws to minimize discomfort.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Andersen, PhD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu